CLINICAL TRIAL: NCT01590719
Title: A Randomized, Phase II, Multicenter, Double-Blind, Placebo-Controlled Study Evaluating The Efficacy And Safety Of Onartuzumab (MetMAb) In Combination With 5-Fluorouracil, Folinic Acid, And Oxaliplatin (mFOLFOX6) In Patients With Metastatic HER2-Negative Gastroesophageal Cancer
Brief Title: A Study of Onartuzumab (MetMAb) in Combination With mFOLFOX6 in Patients With Metastatic Human Epidermal Growth Factor Receptor 2 (HER2) Negative Gastroesophageal Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: YO28252; 2012-000858-57 (EudraCT Number)
Record Dates: First submitted 2012-05-02; First posted 2012-05-03 (Estimated); Last update posted 2016-08-09 (Estimated); Status verified 2016-08

CONDITIONS: Gastric Cancer
MeSH Terms: conditions — Stomach Neoplasms | interventions — onartuzumab; Oxaliplatin; Leucovorin; Fluorouracil

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Onartuzumab (MetMAb) with mFOLFOX6 (Experimental): Onartuzumab (MetMAb) in combination with mFOLFOX6 (modified 5-fluorouracil, folinic acid [leucovorin], and oxaliplatin)
  Interventions: Drug: Onartuzumab (MetMAb); Drug: Oxaliplatin; Drug: Folinic acid; Drug: Levofolinic acid; Drug: 5-Fluorouracil
- Placebo with mFOLFOX6 (Placebo Comparator): Placebo in combination with mFOLFOX6 (modified 5-fluorouracil, folinic acid [leucovorin], and oxaliplatin)
  Interventions: Drug: Placebo; Drug: Oxaliplatin; Drug: Folinic acid; Drug: Levofolinic acid; Drug: 5-Fluorouracil

INTERVENTIONS:
Drug: Placebo — Repeating intravenous dose until disease progression, unacceptable toxicity, or patient or physician decision to discontinue treatment
  Arms: Placebo with mFOLFOX6
Drug: Onartuzumab (MetMAb) — Repeating intravenous dose until disease progression, unacceptable toxicity, or patient or physician decision to discontinue treatment
  Arms: Onartuzumab (MetMAb) with mFOLFOX6
Drug: Oxaliplatin — Oxaliplatin 85 mg/m2 IV every 2 weeks until disease progression, unacceptable toxicity, or patient or physician decision to discontinue treatment
Drug: Folinic acid — Folinic acid 400 mg/m2 every 2 weeks until disease progression, unacceptable toxicity, or patient or physician decision to discontinue treatment
Drug: Levofolinic acid — If folinic acid is unavailable: levofolinic acid 200 mg/m2 every 2 weeks until disease progression, unacceptable toxicity, or patient or physician decision to discontinue treatment
Drug: 5-Fluorouracil — 5-Fluorouracil 400 mg/m2 IV followed by 2400 mg/m2 IV infusion every 2 weeks until disease progression, unacceptable toxicity, or patient or physician decision to discontinue treatment

SUMMARY:
This randomized, multicenter, double-blind, placebo-controlled study will evaluate the efficacy and safety of onartuzumab (MetMAb) in combination with mFOLFOX6 in patients with metastatic HER2-negative adenocarcinoma of the stomach or gastroesophageal junction. Patients will be randomized in a 1:1 ratio to receive either onartuzumab (MetMAb) or placebo in combination with mFOLFOX6. Patients may continue to receive onartuzumab (MetMAb) or placebo until disease progression, unacceptable toxicity, patient or physician decision to discontinue treatment.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients, 18 years of age and older
* Adenocarcinoma of the stomach or gastroesophageal junction with inoperable, metastatic disease, not amenable for curative therapy
* Eastern Cooperative Oncology Group (ECOG) performance status 0 or 1
* Life expectancy >3 months
* Presence of tissue sample for immunohistochemistry assay of Met receptor and HER2 status (if unknown)
* Radiographic evidence of disease; measurable disease or non-measurable but evaluable disease, according to the Response Evaluation Criteria in Solid Tumors (RECIST v1.1); Patients with peritoneal disease would generally be regarded as having evaluable disease and allowed to enter the trial.
* For women who are not postmenopausal or surgically sterile; agreement to use an adequate method of contraception (e.g., hormonal implant) during the treatment period and for at least 90 days after the last dose of onartuzumab/placebo and 6 months after the last dose of oxaliplatin
* For men: agreement to use a barrier method of contraception during the treatment period and for 90 days after the last dose of onartuzumab/placebo and 6 months after the last dose of oxaliplatin
* Adequate laboratory values

Exclusion Criteria:

* HER2-positive tumor (primary tumor or metastasis)
* Previous chemotherapy for locally advanced or metastatic gastric carcinoma (adjuvant or neoadjuvant chemotherapy must be completed at least 6 months prior to randomization)
* Prior treatment with investigational drugs that target the hepatocyte growth factor (HGF) or Met pathway
* History of other malignancy within the previous 5 years, except for appropriately treated and presumed cured carcinoma in situ of the cervix, non-melanoma skin carcinoma, Stage 1 uterine cancer, and localized prostate cancer
* Receipt of an investigational drug within 28 days prior to study start
* Clinically significant gastrointestinal abnormalities, except from gastric cancer (e.g., Crohn's disease)
* Significant history of cardiac disease
* Significant vascular disease
* Infection with human immunodeficiency virus, hepatitis B, or hepatitis C

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 123 (Actual)
Dates: Start 2012-07; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
Progression-free survival (PFS) in all patients | Up to 18 months
Progression-free survival (PFS) in patients with Met-positive tumors | Up to 18 months

SECONDARY OUTCOMES:
Safety: incidence of adverse events | 18 months
Overall survival (OS) | 18 months
Overall response rate (ORR) | 18 months
Duration of response (DOR) | 18 months

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (30):
- United States (18):
  - Denver, Colorado
  - New Haven, Connecticut
  - Fort Myers, Florida
  - St. Petersburg, Florida
  - Chicago, Illinois
  - Niles, Illinois
  - Albany, New York
  - New York, New York
  - Cincinnati, Ohio
  - Nashville, Tennessee
  - Austin, Texas
  - Bedford, Texas
  - Garland, Texas
  - The Woodlands, Texas
  - Tyler, Texas
  - Fairfax, Virginia
  - Richmond, Virginia
  - Vancouver, Washington
- Australia (6):
  - Sydney, New South Wales
  - Herston, Queensland
  - Woodville South, South Australia
  - East Bentleigh, Victoria
  - Heidelberg, Victoria
  - Nedlands, Western Australia
- Singapore, Singapore
- Seoul, South Korea
- Taiwan (3):
  - Tainan
  - Taipei
  - Taoyuan
- Bangkok, Thailand

REFERENCES:
- [Derived] Shah MA, Cho JY, Tan IB, Tebbutt NC, Yen CJ, Kang A, Shames DS, Bu L, Kang YK. A Randomized Phase II Study of FOLFOX With or Without the MET Inhibitor Onartuzumab in Advanced Adenocarcinoma of the Stomach and Gastroesophageal Junction. Oncologist. 2016 Sep;21(9):1085-90. doi: 10.1634/theoncologist.2016-0038. Epub 2016 Jul 8. PMID 27401892